CLINICAL TRIAL: NCT04798794
Title: Association Between Early Change in PaCO2 After ECMO Initiation and Neurological Outcome in Newborns
Brief Title: PCO2 ELSO (Extracorporeal Life Support Organization)
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JS
Record Dates: First submitted 2021-03-05; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Failure
Keywords: Ecmo; Neonates
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ECMO for neonates — Neonates (<28 j) supported by ECMO for severe respiratory failure

SUMMARY:
Investigation of the association between PaCO2 change after extra corporeal membrane oxygenation (ECMO) initiation and neurological outcome and mortality in neonates treated by ECMO for respiratory failure.

DETAILED DESCRIPTION:
Retrospective analysis of the ELSO database investigating the association between the change of PCO2 value after ECMO start and the risk of acute neurological event under ECMO defined by the onset of cerebral bleeding and/or ischemic stroke and/or clinical or electrical seizure and/or brain death.

ELIGIBILITY:
Inclusion Criteria :

* Support by ECMO for respiratory indication

Exclusion Criteria :

* None

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates (<28 j) supported by ECMO for severe respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 4072 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Acute Neurological Event | Up to 90 days after ECMO initiation
  Onset of cerebral bleeding and/or ischemic stroke and/or clinical or electrical seizure and/or brain death. The outcome (ANE) was defined by the occurrence of almost one of the following item:
  * Ischemic or hemmorrhagic stroke diagnosed by ultrasounds, CT or MRI
  * Clinical or electrical seizures : diagnosed by ElectroEncepahloGraphy (EEG)
  * Brain death clinically diagnosed

SECONDARY OUTCOMES:
28-day mortality | 28 days after ECMO start
  Newborns died after 28 days despite ECMO assistance

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No